CLINICAL TRIAL: NCT00002350
Title: A Phase I Trial of APL 400-003 Vaccine: Safety and Immune Response Evaluations of Multiple Injections at Escalating Doses in Asymptomatic HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apollon (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 089; APL 400-003RX101
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-07

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; AIDS Vaccines; DNA, Viral
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: APL 400-003

SUMMARY:
To evaluate safety and immune response in HIV-infected patients treated with multiple injections of APL 400-003 vaccine.

PER 2/27/96 AMENDMENT: To evaluate the safety of the vaccine when administered via the Biojector 2000 Needle-Free Injection Management System.

Facilitated DNA inoculation, a new type of DNA vaccine, involves direct injection of non-infectious HIV genes into a patient's muscle, along with agents that promote uptake of the genes into host cells. Host cells that have taken up these genes then produce viral proteins in a form that elicits immune responses in the form of antibodies, killer T-cells, and helper T-cells. The safety of this new vaccine approach needs to be assessed.

PER 2/27/96 AMENDMENT: The Biojector 2000 provides an option for delivering the vaccine without a needle and employs a single-use syringe to avoid cross-contamination.

DETAILED DESCRIPTION:
Facilitated DNA inoculation, a new type of DNA vaccine, involves direct injection of non-infectious HIV genes into a patient's muscle, along with agents that promote uptake of the genes into host cells. Host cells that have taken up these genes then produce viral proteins in a form that elicits immune responses in the form of antibodies, killer T-cells, and helper T-cells. The safety of this new vaccine approach needs to be assessed.

PER 2/27/96 AMENDMENT: The Biojector 2000 provides an option for delivering the vaccine without a needle and employs a single-use syringe to avoid cross-contamination.

Patients are given intramuscular injections of APL 400-003 at one of three doses (30, 100, or 300 mcg) on day 0 and again at weeks 10 and 20, and followed for 16 weeks after the final dose. An 8-week period prior to initial dosing is required for immortalizing the patient's PBMCs.

PER 2/27/96 AMENDMENT: Five patients will be evaluated at the 300 mcg dose with the Biojector 2000.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Low doses of nonprescription NSAIDS, acetaminophen, ibuprofen, aspirin, replacement hormone therapy, and vitamin supplements.

Patients must have:

* Asymptomatic HIV infection with no acute related infection.
* CD4 count >= 500 cells/mm3.
* Normal hematologic, renal, hepatic, metabolic, and endocrine function.

NOTE:

* No more than one patient over 50 years of age is permitted at each dose level.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Residual toxicity from prior drug treatment.
* Hypersensitivity to bupivacaine or amide-type local anesthetic.
* Active viral hepatitis, autoimmune disorders, or other debilitating chronic diseases.

Concurrent Medication:

Excluded:

* Medications that affect immune function.
* Antiretrovirals.

Patients with the following prior conditions are excluded:

* Malignancies other than curatively treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* History of anaphylaxis to vaccines.

Prior Medication:

Excluded:

* Prior immunization with any experimental HIV vaccines.
* Other experimental therapy within 30 days prior to study entry.
* Prior cancer chemotherapy.
* Antiretrovirals within 3 months prior to study entry.

Prior Treatment:

Excluded:

* Prior radiotherapy. IV drug use or any other high-risk behavior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16

CONTACTS AND LOCATIONS:
Locations (1):
- Univ of Pennsylvania Med Ctr, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] MacGregor RR, Gluckman S, Lacy K, Kaniefski B, Boyer J, Wang B, Bagarazzi M, William WV, Francher D, Ginsberg R, Higgins T, Weiner D. First human trial of a facilitated DNA plasmid vaccine for HIV-1: safety and host response. Int Conf AIDS. 1996 Jul 7-12;11(2):23 (abstract no WeB293)
- [Background] MacGregor R, Gluckman S, Lacy K, Wang B, Ugen K, Chattergoon M, Bagarazzi J, Williams W, Ginsberg R, Higgins T, Boyer J, Weiner D. A DNA plasmid vaccine for HIV-1: experience in the first human trial indicates humoral and cell-immune responses. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:142 (abstract no 421)